CLINICAL TRIAL: NCT04668521
Title: Multifactorial Risk Assessment for Breast & Ovarian Cancer Risk Detection
Acronym: OVA360
Status: Terminated | Type: Observational
Why Stopped: cohort C looked at feasibility of genetics & protein to evaluate risk with a family hx of cancer or associated variant. Since few patients show these factors, this approach would not yield sufficient information to make inferences
Sponsor: Aspira Women's Health (Industry)
Responsible Party: Sponsor
Other Study IDs: 05-2019
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Adnexal Mass; Germline BRCA1 Gene Mutation; Germline BRCA2 Gene Mutation; Hereditary Breast and Ovarian Cancer
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COHORT A: Women with a pelvic mass, symptomatic or asymptomatic.
  Interventions: Other: OVA360
- COHORT B: Women diagnosed with a pelvis mass undergoing genetic testing through our commercial offering.
  Interventions: Other: OVA360
- COHORT C: Subject must not have an identifiable adnexal mass and may, or may not, have a family history or a known familial genetic abnormality (germ line or identified in family cancer i.e. somatic DNA mutation) associated with ovarian cancer.
  Interventions: Other: OVA360

INTERVENTIONS:
Other: OVA360 — Multifactorial Risk Assessment for Breast & Ovarian Cancer Risk Detection

SUMMARY:
The objective of this project is to validate a next-generation assay that utilizes both the protein biomarkers of our already established ovarian cancer risk assessment combined with a molecular profile in both germline and early somatic detection.

ELIGIBILITY:
Key inclusion criteria:

* Female subject
* 18 years of age or older

Cohort A specific inclusion criteria:

• Diagnosed with a pelvic mass

Cohort B specific inclusion criteria:

* Diagnosed with a pelvic mass
* Undergoing genetic testing through our commercial offering

Cohort C specific inclusion criteria:

• Subject must not have an identifiable adnexal mass and may, or may not, have a family history or a known familial genetic abnormality (germ line or identified in family cancer i.e. somatic DNA mutation) associated with ovarian cancer.

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with or without a pelvic mass.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
OVA360 | 12 months
  Identify the molecular key driver of Ovarian cancer and develop a diagnostic test for early Ovarian cancer detection

CONTACTS AND LOCATIONS:
Overall Officials: Todd Pappas, PhD, Principal Investigator — Aspira Women's Health
Locations (1):
- Silvana Franco, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No